CLINICAL TRIAL: NCT00339794
Title: Clinical Integration of Genetic Risk Assessment in Family Medicine
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905055; 05-HG-N055
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-16

CONDITIONS: Genomics
Keywords: Racial Profiling; Genomics; Genetic Testing; Family History; Family Physician

SUMMARY:
This study, conducted by the American Academy of Family Physicians (AAFP) and the National Human Genome Research Institute, will characterize family physicians' attitudes and practices related to the genetics of complex disorders. As the front line of care for most Americans, family medicine will have a central role in seeing that new findings in genetics lead to disease prevention and health improvements. The information gained from this study could be useful in understanding and shaping the dissemination of genetic medicine in ways that improve the standard of primary care practice.

Members of the AAFP will be randomly selected from the organization's membership records to be invited to participate in this two-phase study. The first phase is a web-based survey of AAFP members. In the second phase, a sub-sample of those who complete the survey will be re-contacted; half will be members who have enrolled in a year-long web-based curriculum related to medical genetics, and the other half will be those who have chosen not to enroll in the curriculum.

Survey questions relate to the physicians' practices, knowledge, and opinions about implications of genomic medicine. Survey areas include family history taking; opinions about the future of genetics and family medicine; information about the physician and his or her practice; and physician's skills, attitudes and knowledge.

DETAILED DESCRIPTION:
Although the evidence base for genetic susceptibility markers for complex disorders (e.g., diabetes, hypertension, and obesity) and the clinical utility of the related genetic tests has not been demonstrated, all signs suggest that genetics will become increasingly relevant to and integrated into family medicine. In recognition of these emerging genomic innovations and their potential for improving primary care practice, the American Academy of Family Physicians (AAFP), in collaboration with the National Human Genome Research Institute (NHGRI), has made genomic medicine the topic of their 2005 Annual Clinical Focus curriculum. The AAFP is one of the largest medical organizations with a membership that comprises a group of 56,400 active family physicians who deliver care in a broad array of practice settings in rural and urban communities around the United States, Puerto Rico, the Virgin Islands and Guam. This study seeks to take advantage of the plans for AAFP's clinical focus on genomics to characterize family physicians' attitudes and practices related to the genetics of complex disorders. This information could be useful in understanding and shaping the dissemination of genetic medicine in ways that improve the standard of primary care practice. To this end, we propose to conduct two phases of research activity. In the first phase, a web-based survey will be conducted of members of AAFP. In the second phase, a sub-sample of those who complete the survey will be re-contacted; half will be members who have enrolled in a year-long web-based curriculum related to medical genetics, and the other half will be those who have chosen not to enroll in the curriculum.

ELIGIBILITY:
* INCLUSION CRITERIA:

The sampling frame for this study is the American Academy of Family Physicians (AAFP) membership (estimated at 54,600 active members). The majority of the members of AAFP are physicians with a family physicians residency background (89%) who tend to practice in urban (71%), private office settings (89%) and provide direct patient care (82%).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2004-12-07; Study Completion 2010-07-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sayers MD, Bellack AS, Wade JH, Bennett ME, Fong P. An empirical method for assessing social problem solving in schizophrenia. Behav Modif. 1995 Jul;19(3):267-89. doi: 10.1177/01454455950193001. PMID 7625993
- [Background] Burchard EG, Ziv E, Coyle N, Gomez SL, Tang H, Karter AJ, Mountain JL, Perez-Stable EJ, Sheppard D, Risch N. The importance of race and ethnic background in biomedical research and clinical practice. N Engl J Med. 2003 Mar 20;348(12):1170-5. doi: 10.1056/NEJMsb025007. No abstract available. PMID 12646676
- [Background] Burke W. Genetic testing. N Engl J Med. 2002 Dec 5;347(23):1867-75. doi: 10.1056/NEJMoa012113. No abstract available. PMID 12466512